CLINICAL TRIAL: NCT04770298
Title: The Effectiveness of the Bobath Neurodevelopmental Treatment and Halliwick Concept Hydrotherapy in the Treatment of Children With Cerebral Palsy.
Brief Title: Effectiveness of Bobath/Halliwick on Children With Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Chandolias, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14018003112
Record Dates: First submitted 2021-02-20; First posted 2021-02-25 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: aquatic therapy; pediatrics; cerebral palsy; Bobath; Halliwick
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 3 groups, 80 children with CP
  1. group: Intervention in water- halliwick, 40 children
  2. group: On land therapy- bobath, 40 children
  3. group: No intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Halliwick Assessment Group (Experimental): 8 children with GROSS MOTOR FUNCTION CLASSIFICATION SYSTEM (GMFCS) I, 13 children with GMFCS II, 7 GMFCS III children, 8 GMFCS IV children and 4 children with GMFCS V. Intervention in water environment (Halliwick Concept), 1 times/week- 1 intervention on land/week, 9 months duration.
  Interventions: Other: Halliwick Concept
- Bobath Assessment Group (Experimental): 7 children with GMFCS I, 12 children with GMFCS II, 8 children with GMFCS III, 6 children with GMFCS IV and 2 children with GMFCS V. Intervention on land ( Bobath), 2 times/week, 9 months duration.
  Interventions: Other: Halliwick Concept
- No intervention group (No Intervention): 1 children with GMFCS I, 1 child with GMFCS III, 1 child with GMFCS IV and 2 GMFCS V children. No intervention.

INTERVENTIONS:
Other: Halliwick Concept — Halliwick Concept: Water intervention Bobath Concept: Neurodevelopmental Treatment
  Other Names: Bobath Concept
  Arms: Bobath Assessment Group; Halliwick Assessment Group

SUMMARY:
Investigation of the effectiveness of water based therapy on children with Cerebral Palsy (CP)

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial was:

To examine the effectiveness of the Halliwick concept intervention in water approach for people with motor deficiency and, more specifically, for children with diagnosed cerebral palsy.

In a second phase, to compare the contribution of water intervention to the child's motor development against just Bobath physiotherapeutic intervention, in terms of the milestones of gross motor skills of the children over time.

The aim of the research is to determine the contribution of the Halliwick Concept- Hydrotherapeutic Intervention approach in the psychomotor development in children with cerebral palsy and to explore its contribution to a comprehensive therapeutic approach for these children. It is a fact that, in recent years, parallel therapeutic approaches have gained ground, which, in combination with the physiotherapeutic treatment, contributes to the enhancement of therapeutic effects in early and follow-up intervention for children with cerebral palsy.

The study resulted from the fact that there is not such a large-scale study in Greece. Also, there are few published studies in the world, trying to evaluate the therapeutic benefit of the Halliwick Concept as an hydro-therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy
* Not have some type of surgery or botulinum toxin infusion in the last year.
* The children with cognitive limitations were selected, in order to be able to execute elementary commands.
* Attending treatment program by the same therapist, either on water, or on land.

Exclusion Criteria:

* Children with autism
* Children who had some scheduled surgery or botulinum toxin injection.
* Children with severe vision problems
* Children who could not follow the verbal instructions or reproduce a test reproduction.
* Children who were absent from the treatment program either in the water or on land for over a week

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-26 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
GMFM | 9 months
  GROSS MOTOR FUNCTION MEASURE (Scale for gross mobility) (scoring 0%-100%)
PEDI | 9 months
  PEDIATRIC EVALUATION OF DISABILITY INVENTORY (Scale for assess the daily life activities) (scoring 0%-100%)
PBS | 9 months
  PAEDIATRIC BALANCE SCALE (BERG BALANNCE SCALE MODIFIED) (Scale for assess the balance) (score 0-56)
TUG | 9 months
  TIMED UP AND GO (Scale to asses speed) (the minimoum time the better)
WOTA 1 | 9 MONTHS
  WATER ORIENTATION TEST ALYN 1 (Aquatic Scale to asses adaptation in water environment) (Aquatic Score 0- 52)
WOTA 2 | 9 months
  WATER ORIENTATION TEST ALYN 12 (Aquatic Scale to asses adaptation in water environment) ( Score 0-81)
SWIM | 9 months
  SWIM WITH INDEPENDENT MEASURE (Aquatic Scale to asses adaptation in water environment) (Score 0-71)
HAAR | 9 months
  HUMPHRIES' ASSESSMENT OF AQUATIC READINESS (Aquatic Scale to asses adaptation in water environment)(Score 0-34)

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Tsiokanos, Dr, Study Director — Univesity of Thessaly
Locations (1):
- University of Thessaly, Lamía, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimitrijevic L, Aleksandrovic M, Madic D, Okicic T, Radovanovic D, Daly D. The effect of aquatic intervention on the gross motor function and aquatic skills in children with cerebral palsy. J Hum Kinet. 2012 May;32:167-74. doi: 10.2478/v10078-012-0033-5. Epub 2012 May 30. PMID 23487257

DOCUMENTS (1):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04770298/Prot_000.pdf